CLINICAL TRIAL: NCT02839278
Title: Biological Evaluation of a Novel Anti-inflammatory Treatment in Immune-mediated Inflammatory Diseases
Acronym: Super-Bio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P/2014/233
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Inflammation
Keywords: Immunomodulation
MeSH Terms: conditions — Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immune-mediated inflammatory disease (Experimental): Patients with an immune-mediated inflammatory disease. A blood sample is achieved at T0 (no follow-up).
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample

SUMMARY:
The aim of the study is to investigate in vitro the impact of a novel anti-inflammatory treatment on costimulatory molecules expressed on monocytes.

ELIGIBILITY:
Inclusion Criteria:

* Immune-mediated inflammatory disease (non-ST segment elevation myocardial infarction, Rheumatoid arthritis, Chronic obstructive pulmonary disease, Idiopathic pulmonary fibrosis, Crohn's disease, Ulcerative colitis, Cystic fibrosis, Psoriasis, Multiple sclerosis or major depressive episode)
* Patient able to understand the reason of the study
* Patient not opposed to the conservation of biological samples for scientific research

Exclusion Criteria:

* Pregnant woman
* Subject without health insurance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-04; Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Expression of costimulatory molecules CD86, CD80, CD40 and class II (HLA-DR) on monocytes | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No